CLINICAL TRIAL: NCT01006538
Title: A Randomised Controlled Trial of Epimacular Brachytherapy Versus Ranibizumab Monotherapy for the Treatment of Subfoveal Choroidal Neovascularisation Associated With Wet Age-related Macular Degeneration in Patients Who Have Commenced Anti-VEGF Therapy
Brief Title: Macular EpiRetinal Brachytherapy Versus Lucentis® Only Treatment (MERLOT)
Acronym: MERLOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09/HO206/20; 2009-012509-20 (EudraCT Number)
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2019-05

CONDITIONS: Macular Degeneration
Keywords: Wet Age-related Macular Degeneration; Predominantly classic; Minimally classic; Occult with no classic; Retinal Angiomatous Proliferation (RAP) lesions
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (treatment) (Experimental): Arm A: A single surgical procedure with epimacular brachytherapy using the VIDION® System, with Lucentis® (0.5 mg) administered on a monthly basis as required.
  Interventions: Device: Epimacular Brachytherapy; Drug: Ranibizumab
- Arm B (control): (Active Comparator): Arm B: Lucentis® (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria below.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Device: Epimacular Brachytherapy — Strontium-90. The device delivers 24 Gray of beta radiation to the choroidal neovascular membrane (CNV) lesion. Each device is calibrated for a set duration.
  Other Names: Vidion System; EpiRetinal Brachytherapy
  Arms: Arm A (treatment)
Drug: Ranibizumab — intravitreal injection of Ranibizumab (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria
  Other Names: Lucentis; Anti-VEGF therapy

SUMMARY:
Wet age-related macular degeneration is the most common cause of blind registration in the United Kingdom (UK). Standard treatment involves regular eye injections of a drug called ranibizumab (Lucentis). For most patients, ranibizumab maintains their vision but the effect of the drug is temporary, and they therefore require monthly hospital visits and typically six injections into the eye every year, probably for life.

This study tests a new surgical device that delivers a focal dose of radiation (epimacular brachytherapy) to the macula (the part inside the back of the eye that gives fine central vision), to try and reduce or eliminate the need for ongoing, regular eye injections. The trial compares epimacular brachytherapy to ongoing standard treatment with ranibizumab.

Whereas most studies of this new surgical device target patients who have not yet commenced any treatment, this study targets those who are requiring frequent eye injections, as there are limited surgical resources and these resources are best directed to those who have not fully responded to ranibizumab therapy, or whose response is shortlived. These patients have the most to gain from a device that may reduce their burden of treatment. The findings in untreated disease cannot be extrapolated to this discrete subset of patients, hence the need for a study that targets refractory disease.

It is hypothesised that epimacular brachytherapy will reduce the frequency of Lucentis® (ranibizumab) re-treatment that patients require, whilst maintaining visual acuity.

DETAILED DESCRIPTION:
The eye is designed like a camera, with a lens at the front and a film at the back. Using this analogy, the retina is the film in the camera. In the center of the retina is the macula, the region that absorbs focused light from the lens and creates an image of the outside world that is then transmitted to the brain.

The commonest cause of irreversible blindness in developed nations is age related macular degeneration (AMD). There are two types, 'dry' and 'wet' AMD. Wet AMD is also called neovascular AMD: It is the most damaging type and can blind people in a matter of weeks. Neovascular AMD is due to the growth of blood vessels under the retina, similar to a wound healing process. The blood vessels grow in two patterns, classic (15%) and occult (85%); these can be visualized with fluorescein angiography, a commonly used technique that photographs the macula after a fluorescent dye is injected into the arm. In most research on AMD, vision is assessed using the Early Treatment of Diabetic Retinopathy Study (ETDRS) vision chart, with results quantified in numbers of letters read correctly, from 0 (very poor vision) to 100 (very good vision).

A new treatment has recently been licensed in the UK called ranibizumab (trade name, Lucentis). This is an antibody that reduces the effect of vascular endothelial growth factor (VEGF), a chemical that mediates new blood vessel growth. This drug is injected into the eye at regular intervals (up to 12 a year, and typically 6 a year). Patients receiving 12 ranibizumab injections per year have a greater than 90% chance of maintaining their vision over 12 months (1-2). Another drug called bevacizumab (Avastin) has been used off label (without a licence) in the UK, USA and other countries, and this also targets VEGF. In non-randomized trials it showed similar results to ranibizumab, and is currently being assessed in head-to-head trials with ranibizumab in the UK and the USA.

One of the drawbacks of ranibizumab therapy is that patients require regular injections into the eye. In the UK, the National Institute for Health and Care Excellence (NICE) recommends patient with newly diagnosed wet AMD receive three consecutive monthly injections of ranibizumab, followed by 'as required' therapy based on disease activity. They estimate that patients receive eight injections in the first year, six in the second, and ongoing treatment thereafter. Patients require monthly hospital visits for life and each injection caries a small but cumulative risk of complications such as bleeding inside the eye, infection, detachment of the retina, raised eye pressure, and systemic effects such as stroke. A treatment that produced a more durable reduction in disease activity might reduce these risks, be more cost effective for the health service, and reduce the considerable burden of treatment for patients and their carers, with the prospect of fewer hospital visits. It would also give patients an alternative choice, should they not wish to undergo such regular eye injections.

Radiation has the potential to produce a more durable therapeutic effect, by targeting the proliferating cells that cause visual damage in wet AMD. It is well known that radiation can modify the wound healing process, which is a biological process similar to neovascular AMD. Previous studies with external beam radiation have shown an effect on the progression of macular degeneration. However vision was not improved - possibly due to the type of radiation used, the accuracy of delivery, and collateral damage to neighbouring structures.

Epimacular brachytherapy delivers local, controlled radiation 1-3 mm into the macula, during an operation called a vitrectomy. The proposed device will be CE marked (Conformité Européene - approved for clinical use) and is manufactured by NeoVista Inc, who have completed preliminary trials to assess the safety and feasibility of treating naive (newly diagnosed) neovascular AMD with a single application of brachytherapy. Initial data showed that epiretinal treatment stabilised vision for most patients with neovascular AMD. Phase II trials using the device with two concomitant doses of bevacizumab showed promising results with 91% of patients maintaining vision (losing fewer than 15 ETDRS letters), with an average improvement of 8.9 ETDRS letters (3). The percentage of patients whose visual acuity improved by more than 3 lines (15 letters on the ETDRS scale) was 38%. These results are similar to the large studies of monthly ranibizumab. A mean gain of 8.9 letters is more than twice the visual gain reported in large studies (HORIZON) of 'as required' dosing, as occurs in the UK.

A large, international, randomized, multicentre study of the device, used with two concomitant injections of ranibizumab, is now underway (the CABERNET study). Recruitment is occuring in the hospital of the applicant, and two other UK sites, with more sites to follow. The CABERNET study uses the device in treatment naive disease and was favourably reviewed by the Southwest Research Ethics Committee (07/H0206/50).

Whilst the CABERNET study will provide high quality data in treatment naive disease, it is not possible to rely on this study in relation to previously treated disease. Prior therapy with ranibizumab modifies the disease process, and those that respond poorly to injections differ from the majority, suggesting differences in the underlying disease process. It is therefore necessary to study the subset of patients with refractory disease, if valid clinical conclusions are to be reached. Furthermore, because there is limited vitreoretinal surgical capacity it is logical to offer surgical intervention to patients who have not responded fully to ranibizumab, rather than aim to treat all patients presenting with wet-AMD. To this end, an uncontrolled study (MERITAGE) using the device in refractory, previously treated disease has commenced, having received a favourable opinion from the Southwest Research Ethics Committee (07/H0206/55). The present randomised controlled trial (MERLOT) follows on from the Phase II MERITAGE study. It targets previously treated disease, and patients that are receiving regular ranibizumab, to determine if the device benefits this large subset of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with subfoveal choroidal neovascularisation associated with wet age-related macular degeneration. Retinal Angiomatous Proliferation (RAP) lesions not directly involving the fovea must be associated with contiguous foveal leakage demonstrated on fundus examination, optical coherence tomography (OCT), or fluorescein angiography;
2. Subjects must have received anti-VEGF induction treatment, defined as the first three months of anti-VEGF therapy. Following this induction period, subjects must have received at least 4 additional injections of Lucentis® in no more than 12 months preceding enrolment, or 2 additional injections of Lucentis® in no more than 6 months preceding enrolment, given on an as needed basis;
3. At the time subjects commenced anti-VEGF therapy for wet age-related macular degeneration they were aged 50 years or older and met the NICE treatment criteria for Lucentis® therapy, as outlined in the Final Appraisal Determination (FAD). This states that all of the following circumstances must apply in the eye to be treated:

   * the best-corrected visual acuity is between 6/12 and 6/96 (24 to 69 ETDRS letters)
   * there is no permanent structural damage to the central fovea
   * the lesion size is less than or equal to 12 disc areas in greatest linear dimension
   * there is evidence of recent presumed disease progression (blood vessel growth, as indicated by fluorescein angiography, or recent visual acuity changes)

Exclusion Criteria:

1. Patients who have not been treated in accordance with NICE guidance;
2. Visual acuity worse than 6/96 at the time of study enrolment;
3. Subjects with prior or concurrent subfoveal CNV therapy with agents, surgery or devices (other than Macugen®, Avastin®, or Lucentis®) including thermal laser photocoagulation (with or without photographic evidence), photodynamic therapy, intravitreal or subretinal steroids, and transpupillary thermotherapy (TTT);
4. Subfoveal scarring;
5. Subjects with active concomitant disease in the study eye, including uveitis, presence of pigment epithelial tears or rips, acute ocular or periocular infection;
6. Subjects who have been previously diagnosed with Type 1 or Type 2 Diabetes Mellitus. Subjects who do not have a documented diagnosis, but have retinal findings consistent with Type 1 or Type 2 Diabetes Mellitus;
7. Subjects with advanced glaucoma (greater than 0.8 cup:disk) or intraocular pressure ≥ 30 mmHg in the study eye;
8. Previous glaucoma filtering surgery in the study eye;
9. Subjects with inadequate pupillary dilation or significant media opacities in the study eye, including cataract, which may interfere with visual acuity or the evaluation of the posterior segment;
10. Current vitreous haemorrhage in the study eye;
11. History of rhegmatogenous retinal detachment or macular hole in the study eye;
12. Subjects who present with CNV due to causes other than AMD, including subjects with known or suspected idiopathic polypoidal choroidal vasculopathy (IPCV), ocular histoplasmosis syndrome, angioid streaks, multifocal choroiditis, choroidal rupture, or pathologic myopia (spherical equivalent ≥ 8 Dioptre or axial length ≥ 25mm);
13. Subjects who have undergone any intraocular surgery in the study eye within 12 weeks prior to the screening visit, with the exception of cataract surgery as discussed in the Exclusion Criteria #14
14. Previous cataract surgery within 2 months prior to enrolment into the study;
15. Subjects with known serious allergies to fluorescein dye used in angiography;
16. Subjects with known sensitivity or allergy to Lucentis®;
17. Subjects who underwent previous radiation therapy to the eye, head or neck;
18. Subjects with an intravitreal device or drug in the study eye;
19. Subjects with any other condition, which in the judgment of the investigator would prevent the subject from completing the study (e.g. documented diagnosis of dementia or serious mental illness);
20. Current participation in another drug or device clinical trial, or participation in such a clinical trial within the last year;
21. History of use of drugs with known retinal toxicity, including: chloroquine (Aralen - an anti-malarial drug), hydroxychloroquine (Plaquenil), phenothiazines, chlorpromazine (Thorazine), thioridazine (Mellaril), fluphenazine (Prolixin), perphenazine (Trilafon), and trifluoperazine (Stelazine);
22. Subjects who are unwilling or unable to return for scheduled treatment and follow-up examinations for three years;
23. Women must be post-menopausal more than 1 year unless surgically sterilised

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2009-11; Primary Completion 2015-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Jackson, PhD FRCOphth, Principal Investigator — King's College Hospital NHS Trust
Locations (24):
- United Kingdom (24):
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Plymouth Royal Eye Infirmary, Plymouth, Devon
  - Torbay Hospital, Torquay, Devon
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Sussex Eye Hospital, Brighton, East Sussex
  - Hull and East Yorks Hospital, Hull, East Yorkshire
  - Essex County Hospital, Colchester, Essex
  - Southend Hospital, Westcliff-on-Sea, Essex
  - Manchester Royal Eye Hospital, Manchester, Greater Manchester
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Maidstone Hospital, Maidstone, Kent
  - Ashford William Harvey Hospital, Willesborough, Kent
  - Royal Liverpool Hospital, Liverpool, Merseyside
  - Arrowe Park Hospital, Upton, Merseyside
  - James Cook Hospital, Middlesbrough, North Yorkshire
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Southampton Hospital, Shirley, Southampton
  - Royal Victoria Infirmary, Newcastle, Tyne and Wear
  - Sunderland Eye Infimary, Sunderland, Tyne and Wear
  - Warwick Hospital Eye Unit, Warwick, Warwickshire
  - St James University Hospital, Leeds, West Yorkshire
  - Bristol Eye Hospital, Bristol
  - Darlington Memorial Hospital, Darlington
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson TL, Soare C, Petrarca C, Simpson A, Neffendorf JE, Petrarca R, Muldrew KA, Peto T, Chakravarthy U, Membrey L, Haynes R, Costen M, Steel DHW, Desai R; MERLOT Study Group. Epimacular brachytherapy for previously treated neovascular age-related macular degeneration: month 36 results of the MERLOT randomised controlled trial. Br J Ophthalmol. 2023 Jul;107(7):987-992. doi: 10.1136/bjophthalmol-2021-320620. Epub 2022 Feb 25. PMID 35217515
- [Derived] Evans JR, Igwe C, Jackson TL, Chong V. Radiotherapy for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 Aug 26;8(8):CD004004. doi: 10.1002/14651858.CD004004.pub4. PMID 32844399
- [Derived] Jackson TL, Soare C, Petrarca C, Simpson A, Neffendorf JE, Petrarca R, Muldrew A, Peto T, Chakravarthy U, Membrey L, Haynes R, Costen M, Steel D, Desai R; MERLOT Study Group. Evaluation of Month-24 Efficacy and Safety of Epimacular Brachytherapy for Previously Treated Neovascular Age-Related Macular Degeneration: The MERLOT Randomized Clinical Trial. JAMA Ophthalmol. 2020 Aug 1;138(8):835-842. doi: 10.1001/jamaophthalmol.2020.2309. PMID 32644148
- [Derived] Jackson TL, Dugel PU, Bebchuk JD, Smith KR, Petrarca R, Slakter JS, Jaffe GJ, Nau JA; CABERNET Study Group. Epimacular brachytherapy for neovascular age-related macular degeneration (CABERNET): fluorescein angiography and optical coherence tomography. Ophthalmology. 2013 Aug;120(8):1597-603. doi: 10.1016/j.ophtha.2013.01.074. Epub 2013 Mar 13. PMID 23490325
- See also: MERLOT Study website with information for Patients and Investigators — http://merlotstudy.com
- See also: Website for King's College Hospital (Study Sponsor Site) — http://www.kch.nhs.uk/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Epimacular Bracytherapy + Lucentis®: Arm A: A single surgical procedure with epimacular brachytherapy using the VIDION® System, with Lucentis® (0.5 mg) administered on a monthly basis as required.
  Epimacular Brachytherapy: Strontium-90. The device delivers 24 Gray of beta radiation to the CNV lesion. Each device is calibrated for a set duration.
- Arm B: Lucentis® Only: Arm B: Lucentis® (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria below.
  Ranibizumab: intravitreal injection (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria
Period: Overall Study
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Started | 244 | 119
Completed | 233 | 115
Not Completed | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm A (Treatment): Arm A: A single surgical procedure with epimacular brachytherapy using the VIDION® System, with Lucentis® (0.5 mg) administered on a monthly basis as required.
  Epimacular Brachytherapy: Strontium-90. The device delivers 24 Gray of beta radiation to the CNV lesion. Each device is calibrated for a set duration.
- Arm B (Control):: Arm B: Lucentis® (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria below.
  Ranibizumab: intravitreal injection (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria
- Total: Total of all reporting groups
Arm/Group | Arm A (Treatment) | Arm B (Control): | Total
Number analyzed (Participants) | 244 | 119 | 363
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 28
  >=65 years | 227 | 108 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (7.2) | 75.8 (7.6) | 76.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 62 | 217
  Male | 89 | 57 | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 244 | 119 | 363
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 244 | 119 | 363

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Early Treatment for Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) From Baseline to Month 12
Description: Manifest refraction and BCVA measurements were performed according to the standard procedure originally developed for Early Treatment for Diabetic Retinopathy Study (ETDRS) and adapted for the Age Related Eye Disease Study (AREDS) protocol. Visual acuity testing was measured at a distance of 4 meters and, for subjects with sufficiently reduced vision, at 1 meter. The ETDRS charts consist of 14 lines, each comprising a series of 5 letters of equal difficulty, with standardized spacing between letters and rows (total 70 letters). Minimum is 0 (no letters read at 1 m) and maximum possible is 100 (70 letters read at 4 m + 30). If visual acuity is so poor that the subject cannot read any of the largest letters at 1 meter count fingers (CF), hand movements (HM) and light perception (PL) are tested.
  The mean change in ETDRS BCVA was calculated from baseline to month 12.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Number analyzed (Participants) | 244 | 119
ETDRS Letters | -4.8 (10.8) | -0.9 (9.7)

2. Primary Outcome: Mean Number of Re-treatment Injections of Lucentis® Per Patient, Per Year.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: injections per patient per year
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Number analyzed (Participants) | 244 | 119
injections per patient per year | 4.8 (3.2) | 4.1 (2.4)

3. Secondary Outcome: Percentage of Subjects Losing < 15 ETDRS Letters
Description: Manifest refraction and BCVA measurements were performed according to the standard procedure originally developed for Early Treatment for Diabetic Retinopathy Study (ETDRS) and adapted for the Age Related Eye Disease Study (AREDS) protocol. Visual acuity testing was measured at a distance of 4 meters and, for subjects with sufficiently reduced vision, at 1 meter. The ETDRS charts consist of 14 lines, each comprising a series of 5 letters of equal difficulty, with standardized spacing between letters and rows (total 70 letters). Minimum is 0 (no letters read at 1 m) and maximum possible is 100 (70 letters read at 4 m + 30). If visual acuity is so poor that the subject cannot read any of the largest letters at 1 meter count fingers (CF), hand movements (HM) and light perception (PL) are tested.
  Participants with worsening in BCVA by less than 15 EDTRS letters at month 12 compared with baseline were considered for this outcome measure.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Number analyzed (Participants) | 244 | 119
Participants | 204 | 110

4. Secondary Outcome: Percentage of Subjects Gaining ≥ 0 ETDRS Letters
Description: Manifest refraction and BCVA measurements were performed according to the standard procedure originally developed for Early Treatment for Diabetic Retinopathy Study (ETDRS) and adapted for the Age Related Eye Disease Study (AREDS) protocol. Visual acuity testing was measured at a distance of 4 meters and, for subjects with sufficiently reduced vision, at 1 meter. The ETDRS charts consist of 14 lines, each comprising a series of 5 letters of equal difficulty, with standardized spacing between letters and rows (total 70 letters). Minimum is 0 (no letters read at 1 m) and maximum possible is 100 (70 letters read at 4 m + 30). If visual acuity is so poor that the subject cannot read any of the largest letters at 1 meter count fingers (CF), hand movements (HM) and light perception (PL) are tested.
  Participants with an improvement in BCVA by more than 0 EDTRS letters at month 12 compared with baseline were considered for this outcome measure.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Number analyzed (Participants) | 244 | 119
Participants | 91 | 55

5. Secondary Outcome: Percentage of Subjects Gaining ≥ 15 ETDRS Letters
Description: Manifest refraction and BCVA measurements were performed according to the standard procedure originally developed for Early Treatment for Diabetic Retinopathy Study (ETDRS) and adapted for the Age Related Eye Disease Study (AREDS) protocol. Visual acuity testing was measured at a distance of 4 meters and, for subjects with sufficiently reduced vision, at 1 meter. The ETDRS charts consist of 14 lines, each comprising a series of 5 letters of equal difficulty, with standardized spacing between letters and rows (total 70 letters). Minimum is 0 (no letters read at 1 m) and maximum possible is 100 (70 letters read at 4 m + 30). If visual acuity is so poor that the subject cannot read any of the largest letters at 1 meter count fingers (CF), hand movements (HM) and light perception (PL) are tested.
  Participants with an improvement in BCVA by more than 15 EDTRS letters at month 12 compared with baseline were considered for this outcome measure.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Number analyzed (Participants) | 244 | 119
Participants | 3 | 6

6. Secondary Outcome: Change in Total Lesion Size by Fluorescein Angiography From Baseline to Month 12
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Number analyzed (Participants) | 219 | 110
mm2 | 1.2 (8.3) | 0.4 (7.6)

7. Secondary Outcome: Change in Total Choroidal Neovascular Membrane (CNV) Size by Fluorescein Angiography From Baseline to Month 12
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Number analyzed (Participants) | 219 | 110
mm2 | 0.5 (7.6) | 1.3 (7.0)

8. Secondary Outcome: Foveal Thickness Measured Using Optical Coherence Tomography (OCT) From Baseline to Month 12
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Arm A: Epimacular Bracytherapy + Lucentis® | Arm B: Lucentis® Only
Number analyzed (Participants) | 225 | 111
μm | -1.0 (215) | 15.7 (196)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) are reported between baseline and month 12.
Groups:
- Arm A: Epimacular Brachytherapy + Lucentis®: Arm A: A single surgical procedure with epimacular brachytherapy using the VIDION® System, with Lucentis® (0.5 mg) administered on a monthly basis as required.
  Epimacular Brachytherapy: Strontium-90. The device delivers 24 Gray of beta radiation to the CNV lesion. Each device is calibrated for a set duration.
  Ranibizumab: intravitreal injection of Ranibizumab (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria
- Arm B (Control): Lucentis ® Only: Arm B: Lucentis® (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria below.
  Ranibizumab: intravitreal injection of Ranibizumab (0.5 mg) administered on a monthly basis as required, using the re-treatment criteria
Arm/Group | Arm A: Epimacular Brachytherapy + Lucentis® | Arm B (Control): Lucentis ® Only
All-Cause Mortality (participants affected / at risk) | 3/244 | 5/119
Serious Adverse Events (participants affected / at risk) | 7/244 | 0/119
Other Adverse Events (participants affected / at risk) | 244/244 | 50/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Epimacular Brachytherapy + Lucentis® (N=244) | Arm B (Control): Lucentis ® Only (N=119)
Endophthalmitis (Eye disorders) | 1 (1) | 0
Postoperative uveitis (Eye disorders) | 2 (2) | 0
Retinal detachment (Eye disorders) | 3 (3) | 0
Visual hallucinations (Eye disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Epimacular Brachytherapy + Lucentis® (N=244) | Arm B (Control): Lucentis ® Only (N=119)
Cataract (Eye disorders) | 82 (82) | 11 (11)
Visual acuity reduced (Eye disorders) | 39 (39) | 8 (8)
Ocular Adverse Events in Study Eye (Eye disorders) | 127 (127) | 31 (31)

LIMITATIONS AND CAVEATS:
Radiation-related microvascular retinal changes may occur beyond the 12 month reporting window (three years' follow up is planned)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No